CLINICAL TRIAL: NCT04300569
Title: A Prospective, Non-Interventional Study to Determine Signs and Symptoms That Impact Daily Life of Patients With Irregular Sleep-Wake Rhythm Disorder and Their Caregivers
Brief Title: A Study to Determine the Signs and Symptoms That Impact Daily Life of Participants With Irregular Sleep-Wake Rhythm Disorder
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2006-A001-111
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-03

CONDITIONS: Irregular Sleep Wake Rhythm Disorder
Keywords: Irregular Sleep-Wake Rhythm Disorder; Alzheimer's disease dementia; Vascular dementia; Circadian Rhythm Sleep Disorder
MeSH Terms: conditions — Dementia, Vascular; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients and Caregivers: Overall Population: Overall population of this study will include both patients with ISWRD associated with AD-D, AD-D with CVD, and/or VaD, and care givers of patients. Patients and caregivers will undergo all study procedures. Caregivers may care either for a patients who undergo all study procedure (including interview) as well for patients who do not undergo any study procedures but give consent or assent for the use of their medical records in the study ("non-interviewed patient").
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — No intervention will be administered.

SUMMARY:
The primary purpose of this study is to determine the signs and symptoms of irregular sleep-wake rhythm disorder (ISWRD) that are important to patients and caregivers of patients with Alzheimer's disease dementia (AD-D), AD-D with cerebrovascular disease (CVD), and/or vascular dementia (VaD) and ISWRD, and to draft an instrument or instruments to assess them.

DETAILED DESCRIPTION:
The study is comprised of an interview with patients and caregivers to determine the signs and symptoms of ISWRD that are important to patients and caregivers of patients.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants

1. Age 60 to 90 years at time of informed consent
2. Documentation of diagnosis of AD-D on the basis of the clinical criteria of the National Institute on Aging/Alzheimer's Association (NIA-AA) diagnostic guidelines and/or VaD on the basis of the National Institute of Neurological Disorders and Stroke (NINDS) and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (AIREN) criteria, and AD-D with CVD on the basis of NINDS-AIREN criteria
3. If the Mini Mental State Examination (MMSE) is conducted (mandatory for clinic visits only) or is available within the past 3 months (all patient participants), MMSE 10 to 26. Note: For all patient participants who undergo a clinic visit, an MMSE must be conducted unless this has been assessed within the past 3 months and the score is available. No MMSE will be conducted during telephone visits, but if a recent MMSE is available, that is, within the past 3 months, that MMSE must be assessed for eligibility.
4. Meets criteria for Circadian Rhythm Sleep Disorder, Irregular Sleep-Wake Type (Diagnostic and Statistical Manual of Mental Disorders - 5th edition [DSM-5]) and the 10th revision of the International Classification of Diseases (ICD-10), as follows: Complaint by the patient or caregiver that the patient has difficulty sleeping during the night and/or has excessive daytime sleepiness associated with multiple irregular sleep bouts during a 24-hour period

   1. Frequency of complaint of sleep and wake fragmentation greater than equal to (>=) 3 days per Week
   2. Duration of complaint of sleep and wake fragmentation >=3 Months
5. If currently taking medications that are used to treat behaviors associated with ISWRD, such as antipsychotic medications or trazodone, the dose must be stable for at least 1 Month
6. Has a caregiver who is also a participant in this study and who meets the eligibility criteria below
7. Is able to speak and understand English or Spanish at a level sufficient to participate in the study interviews, according to the investigator's judgement

Caregivers

1. Age 18 years or older at the time of consent
2. Where the patient is not a study participant (that is, is a non-interviewed patient): The caregiver currently lives with a patient who meets the following criteria:

   1. Has a documented diagnosis of AD-D on the basis of the NIA-AA diagnostic guidelines and/or VaD per NINDS-AIREN criteria
   2. Meets criteria for Circadian Rhythm Sleep Disorder, Irregular Sleep-Wake Type (DSM-5) and the 10th revision of the International Classification of Diseases (ICD-10), as follows: Complaint by the patient or caregiver that the patient has difficulty sleeping during the night and/or has excessive daytime sleepiness associated with multiple irregular sleep bouts during a 24-hour period
3. Is able and willing to provide informed consent or assent.
4. If the MMSE is conducted for the non-interviewed patient (mandatory for clinic visits only) or has been assessed during the past 3 months (all non-interviewed patients), MMSE 10 to 26 Note: For all non-interviewed patients who undergo a clinic visit, the MMSE must be checked for eligibility. The MMSE will be conducted at the clinic visit unless this has been assessed within the past 3 months and the score is available. No MMSE will be conducted during telephone visits, but if a recent MMSE is available,that is, within the past 3 months, that MMSE must be assessed for eligibility.)
5. Is sufficiently familiar (as determined by the investigator) with the patient participant or non-interviewed patient to provide accurate data. The caregiver must share the patient's domicile for an average of at least 5 days and 5 overnights per week for at least the past 3 months
6. Able to speak and understand English or Spanish at a level sufficient to participate in the study interviews, according to the investigator's judgement
7. Willing to have the interview audio recorded

Exclusion Criteria:

Patient Participants

1. A diagnosis of a Lewy body dementia (including Parkinson's disease dementia or dementia with Lewy bodies)
2. A diagnosis of moderate or severe obstructive sleep apnea (OSA), or current use of continuous positive airway pressure (CPAP) even if mild OSA, restless legs syndrome or any other disorder except ISWRD that is likely to impact sleep and interfere with the assessment of ISWRD in the opinion of the investigator

Caregivers

1. The person for whom they care is a non-interviewed patient with any of the following:

   1. A diagnosis of OSA, restless legs syndrome or any other disorder except ISWRD that is likely to impact sleep and interfere with the assessment of ISWRD in the opinion of the investigator
   2. A diagnosis of a Lewy body dementia (including Parkinson's disease dementia or dementia with Lewy bodies)
   3. Evidence of current clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) or any psychiatric disorder other than dementia, that in the opinion of the clinic site investigator could interfere with the assessment of ISWRD
   4. History of drug or alcohol dependency or abuse within approximately the last 2 years
2. Psychotic disorder(s) or unstable recurrent affective disorder(s) as evident by use of antipsychotic medications within approximately the last 2 years
3. History of drug or alcohol dependency or abuse within approximately the last 2 years
4. Current regular use (greater than [>]2) times per week) of medication prescribed to treat insomnia (either approved or off-label)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AD-D, AD-D with CVD and/or VaD and ISWRD and caregivers of patients.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Development of Scale for the Assessment of the Signs and Symptoms of Irregular Sleep-wake Rhythm Disorder (ISWRD) Based on Interview Data | Up to approximately 3 weeks
  Development of scale for the assessment of the signs and symptoms of ISWRD based on interview data of participants using ATLAS ti Coding software will be reported. This study will determine the sleep-wake symptoms and signs that are the most relevant and important from the patient and caregiver perspectives.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - ATP Clinical Research, Costa Mesa, California
  - Pacific Research Network Inc, San Diego, California
  - Miami Jewish Health Systems, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Abington Neurologic Associate, Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on the Eisai website http://eisaiclinicaltrials.com/.